CLINICAL TRIAL: NCT04047602
Title: Radiosurgery Dose Reduction for Brain Metastases on Immunotherapy (RADREMI): A Prospective Pilot Study
Acronym: RADREMI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: trial stopped due to low accrual
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Kevin Shiue, MD, Associate Professor of Clinical Radiation Oncology, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAON-IIR-IUSCC-0710
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Brain Tumor; Brain Metastases; Brain Cancer
Keywords: Radiation; Immune therapy; Stereotactic Radiosurgery
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Reduced Dose Stereotactic Radiosurgery (Experimental): Subjects will receive one stereotactic radiosurgery (SRS) treatment at a reduced dose based on the brain tumor size concurrently with their standard of care immunotherapy. Subjects will undergo follow up with clinical exams and brain MRI scans at 1, 3, 6, 9, and 12 months post SRS treatment
  Interventions: Radiation: Reduced Dose SRS

INTERVENTIONS:
Radiation: Reduced Dose SRS — Subjects will receive SRS treatment at a reduced dose based on the brain tumor size

SUMMARY:
This study will evaluate the rate of radiation necrosis following treatment with immune checkpoint inhibitor (ICI) treatment and radiation therapy in subjects with metastatic brain cancer. Subjects will be treated with the standard of care immunotherapy followed by radiation therapy via stereotactic radiosurgery at a reduced dose.

DETAILED DESCRIPTION:
This is a prospective, single arm, pilot study to determine the symptomatic radiation necrosis rate at 6 months utilizing dose-reduced stereotactic radiosurgery with immunotherapy for subjects with a diagnosis of 1-10 brain metastases from MRI and tissue diagnosis of primary malignancy.

Primary end-point is 6 month symptomatic radiation necrosis, defined as a 6-month rate of clinical symptomatology requiring steroid administration (i.e. Decadron) and/or operative intervention concomitant with advanced and routine brain imaging findings consistent with radiation necrosis. Follow-up MRIs will be fused with the planning scan for this assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Brain MRI-confirmed 1-10 solid tumor brain metastases
2. Biopsy-confirmed primary malignancy
3. ds-GPA estimated median survival of at least 6 months, for histologies not included in the ds-GPA, publications or noted online at brainmetgpa.com, the PI will use either published or validated data or their best clinical judgment to determine the patient's expected survival
4. Stereotactic radiosurgery candidate per treating Radiation Oncologist
5. ≥ 18 years old at the time of informed consent
6. Ability to provide written informed consent and HIPAA (Health Insurance Portability and Accountability Act) authorization.
7. ALC > 800/ul (Ku et al., 2010)
8. Patients currently on cytotoxic chemotherapy are eligible
9. Patients receiving ICI up to 30 days prior to delivery of SRS are eligible
10. Patients having undergone operative resection for metastatic brain disease within 30 days of immune checkpoint inhibitor (ICI) administration are eligible.

Exclusion Criteria:

1. Major medical illnesses or psychiatric impairments, which in the investigator's opinion will prevent administration or completion of the protocol therapy and/or interfere with follow-up
2. Patients unable to receive MRI Brain
3. Patients with more than 10 brain metastases on MRI Brain imaging
4. Any lesion > 4 centimeter maximum diameter
5. Total volume of metastatic disease more than 30 cubic centimeters
6. Previous whole brain radiation therapy
7. For Cohort 1: Previous stereotactic radiosurgery where the 50% isodose line overlaps with current treatment field
8. For Cohort 2: Patients whose treatment will have a dose overlap within the target from prior treatments of 20% or greater
9. Already receiving chronic dexamethasone (chronic = > 2 weeks) prior to SRS
10. Not a radiosurgical candidate per Radiation Oncology discretion
11. Existing autoimmune disease
12. Patients who have an unknown primary cancer
13. Histology not amenable for SRS (i.e. lymphoma). (Small Cell Lung Cancer IS amenable.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2024-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Shiue, MD, Principal Investigator — Indiana University
Locations (3):
- United States (3):
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Indiana University Methodist Hospital, Indianapolis, Indiana
  - Oregon Health and Sciences, Portland, Oregon

REFERENCES:
- [Derived] McClelland S 3rd, Lautenschlaeger T, Zang Y, Hanna NH, Shiue K, Kamer AP, Agrawal N, Ellsworth SG, Rhome RM, Watson GA. Radiosurgery dose reduction for brain metastases on immunotherapy (RADREMI): A prospective phase I study protocol. Rep Pract Oncol Radiother. 2020 Jul-Aug;25(4):500-506. doi: 10.1016/j.rpor.2020.04.007. Epub 2020 Apr 23. PMID 32477016

RESULTS

PARTICIPANT FLOW:
Groups:
- Reduced Dose Stereotactic Radiosurgery With Immunotherapy: Subjects will receive one stereotactic radiosurgery (SRS) treatment at a reduced dose based on the brain tumor size concurrently with their standard of care immunotherapy. Subjects will undergo follow up with clinical exams and brain MRI scans at 1, 3, 6, 9, and 12 months post SRS treatment
  Reduced Dose SRS: Subjects will receive SRS treatment at a reduced dose based on the brain tumor size
Period: Overall Study
Arm/Group | Reduced Dose Stereotactic Radiosurgery With Immunotherapy
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Includes the patients who started treatment and completed the required follow-up period for the study's primary outcome.
Arm/Group | Reduced Dose Stereotactic Radiosurgery
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.08 (7.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
Corticosteroid Use at Baseline [Count of Participants; unit: Participants]
  No | 10
  Yes | 2
Diagnosis-Specific Graded Prognostic Assessment (ds-GPA) Median Survival at Baseline [Median (Inter-Quartile Range); unit: years] — ds-GPA values were calculated using brainmetgpa.com. Survival and the factors that predict survival vary by diagnosis and the molecular profile of the patient's tumor.
  years | 11.75 [8.30 to 19.38]
Primary Site of Initial Cancer Diagnosis [Count of Participants; unit: Participants]
  Adrenal Gland | 1
  Brain | 1
  Kidney/Renal Pelvis | 2
  Lung | 6
  Melanoma | 2
Number of Lesions at Baseline [Median (Inter-Quartile Range); unit: lesions] | 1.50 [1.00 to 3.00]

OUTCOME MEASURES:

1. Primary Outcome: Symptomatic Radiation Necrosis Proportion
Description: The observed proportion of evaluable patients with symptomatic radiation necrosis by 6-months. Symptomatic radiation necrosis was defined as the rate of clinical symptomatology requiring steroid administration (i.e. Decadron) and/or operative intervention concomitant with advanced and routine brain imaging findings consistent with radiation necrosis.
Time Frame: 6 months
Population: Includes those patients who were evaluable for the 6-month outcomes.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Reduced Dose Stereotactic Radiosurgery With Immunotherapy
Number analyzed (Participants) | 12
proportion of participants | 0.083 [0.002 to 0.385]
Statistical Analysis 1: Comparison: Reduced Dose Stereotactic Radiosurgery With Immunotherapy; The observed proportion of evaluable patients with symptomatic radiation necrosis was calculated and tested against a baseline 6-month symptomatic radiation necrosis rate of 16% at a type I error rate of 5% using a one-sided binomial exact test. The null hypothesis is that the observed proportion is equivalent to 16% or 0.160; Test type: Equivalence — The observed proportion of evaluable patients with symptomatic radiation necrosis was calculated and tested against a baseline 6-month symptomatic radiation necrosis rate of 16% at a type I error rate of 5% using a one-sided binomial exact test. The null hypothesis is that the observed proportion is equivalent to 16% or 0.160; p = 0.234, Exact Binomial Test — The p-value reported is the one-sided p-value from the exact equivalence binomial test using an alpha value of 0.05; Binomial Proportion = 0.083, 95% CI 2-sided [0.002 to 0.385] — The binomial proportion 95% confidence intervals were calculated using the Clopper-Pearson (Exact) method

2. Secondary Outcome: Symptomatic Radiation Necrosis Rate
Description: Symptomatic radiation necrosis was defined as the rate of clinical symptomatology requiring steroid administration (i.e. Decadron) and/or operative intervention concomitant with advanced and routine brain imaging findings consistent with radiation necrosis. This measure details the estimated 6-month survival and associated 95% confidence interval from the Kaplan Meier method. The time from treatment start to the presence of symptomatic radiation necrosis was calculated. Patients who did not experience the outcome were censored at the date last known alive or at the date of death if they expired.
Time Frame: 6 months
Population: Includes the patients who were evaluable for the 6-month outcomes.
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | Reduced Dose Stereotactic Radiosurgery With Immunotherapy
Number analyzed (Participants) | 12
survival probability | 0.913 [0.524 to 0.987]

3. Secondary Outcome: Symptomatic Radiation Necrosis Rate
Description: Symptomatic radiation necrosis was defined as the rate of clinical symptomatology requiring steroid administration (i.e. Decadron) and/or operative intervention concomitant with advanced and routine brain imaging findings consistent with radiation necrosis. This measure details the estimated 12-month survival and associated 95% confidence interval from the Kaplan Meier method. The time from treatment start to the presence of symptomatic radiation necrosis was calculated. Patients who did not experience the outcome were censored at the date last known alive or at the date of death if they expired.
Time Frame: 12 months
Population: Includes the patients who were evaluable for the 12-month outcomes.
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | Reduced Dose Stereotactic Radiosurgery With Immunotherapy
Number analyzed (Participants) | 12
survival probability | 0.913 [0.524 to 0.987]

4. Secondary Outcome: Symptomatic Radiation Necrosis by SRS Group
Description: as for outcome 3
Time Frame: 12 months
Population: Includes the patients who were evaluable for the 12-month outcomes.
Measure: Number (95% Confidence Interval); unit: survival probability
Groups:
- Gamma Knife: Subjects received Gamma Knife SRS.
  Subjects will receive one stereotactic radiosurgery (SRS) treatment at a reduced dose based on the brain tumor size concurrently with their standard of care immunotherapy. Subjects will undergo follow up with clinical exams and brain MRI scans at 1, 3, 6, 9, and 12 months post SRS treatment
  Reduced Dose SRS: Subjects will receive SRS treatment at a reduced dose based on the brain tumor size
- Linear Accelerator: Subjects received Linear Accelerator SRS.
  Subjects will receive one stereotactic radiosurgery (SRS) treatment at a reduced dose based on the brain tumor size concurrently with their standard of care immunotherapy. Subjects will undergo follow up with clinical exams and brain MRI scans at 1, 3, 6, 9, and 12 months post SRS treatment
  Reduced Dose SRS: Subjects will receive SRS treatment at a reduced dose based on the brain tumor size
Arm/Group | Gamma Knife | Linear Accelerator
Number analyzed (Participants) | 8 | 4
survival probability | 0.875 [0.387 to 0.981] | 1.000 [1.000 to 1.000]
Statistical Analysis 1: Comparison: Gamma Knife vs Linear Accelerator; The method of Klein et al., (Klein et.al., 2007) was used to compare the 12-month survival probabilities across SRS groups. The null hypothesis was that the survival probabilities were equal; Test type: Other; p = 0.285, Klein Method

5. Secondary Outcome: Symptomatic Radiation Necrosis by Brain Metastases Group
Description: as for outcome 3
Time Frame: 12 months
Population: Includes the patients who were evaluable for the 12-month outcomes.
Measure: Number (95% Confidence Interval); unit: survival probability
Groups:
- Melanoma Brain Metastases: Subjects had melanoma brain metastases at baseline.
  Subjects will receive one stereotactic radiosurgery (SRS) treatment at a reduced dose based on the brain tumor size concurrently with their standard of care immunotherapy. Subjects will undergo follow up with clinical exams and brain MRI scans at 1, 3, 6, 9, and 12 months post SRS treatment
  Reduced Dose SRS: Subjects will receive SRS treatment at a reduced dose based on the brain tumor size.
- Non-Melanoma Brain Metastases: Subjects had non-melanoma brain metastases at baseline.
  Subjects will receive one stereotactic radiosurgery (SRS) treatment at a reduced dose based on the brain tumor size concurrently with their standard of care immunotherapy. Subjects will undergo follow up with clinical exams and brain MRI scans at 1, 3, 6, 9, and 12 months post SRS treatment
  Reduced Dose SRS: Subjects will receive SRS treatment at a reduced dose based on the brain tumor size.
Arm/Group | Melanoma Brain Metastases | Non-Melanoma Brain Metastases
Number analyzed (Participants) | 2 | 10
survival probability | 1.000 [1.000 to 1.000] | 0.900 [0.473 to 0.985]
Statistical Analysis 1: Comparison: Melanoma Brain Metastases vs Non-Melanoma Brain Metastases; The method of Klein et al., (Klein et.al., 2007) was used to compare the 12-month survival probabilities across brain metastases groups. The null hypothesis was that the survival probabilities were equal; Test type: Other; p = 0.292, Klein Method

6. Secondary Outcome: Symptomatic Radiation Necrosis by Immune Checkpoint Inhibitor (ICI) Group
Description: Symptomatic radiation necrosis was defined as the rate of clinical symptomatology requiring steroid administration (i.e. Decadron) and/or operative intervention concomitant with advanced and routine brain imaging findings consistent with radiation necrosis. This measure details the estimated 12-month survival and associated 95% confidence interval from the Kaplan Meier method. The time from treatment start to the presence of symptomatic radiation necrosis was calculated. Ppatients who did not experience the outcome were censored at the date last known alive or at the date of death if they expired.
Time Frame: 12 months
Population: Includes the patients who were evaluable for the 12-month outcomes.
Measure: Number (95% Confidence Interval); unit: survival probability
Groups:
- Single-Agent ICI: Subjects were on a single-agent ICI at baseline.
  Subjects will receive one stereotactic radiosurgery (SRS) treatment at a reduced dose based on the brain tumor size concurrently with their standard of care immunotherapy. Subjects will undergo follow up with clinical exams and brain MRI scans at 1, 3, 6, 9, and 12 months post SRS treatment
  Reduced Dose SRS: Subjects will receive SRS treatment at a reduced dose based on the brain tumor size
- Multi-Agent ICI: Subjects were on a multi-agent ICI at baseline.
  Subjects will receive one stereotactic radiosurgery (SRS) treatment at a reduced dose based on the brain tumor size concurrently with their standard of care immunotherapy. Subjects will undergo follow up with clinical exams and brain MRI scans at 1, 3, 6, 9, and 12 months post SRS treatment
  Reduced Dose SRS: Subjects will receive SRS treatment at a reduced dose based on the brain tumor size
Arm/Group | Single-Agent ICI | Multi-Agent ICI
Number analyzed (Participants) | 9 | 3
survival probability | 0.889 [0.433 to 0.984] | 1.000 [1.000 to 1.000]
Statistical Analysis 1: Comparison: Single-Agent ICI vs Multi-Agent ICI; The method of Klein et al., (Klein et.al., 2007) was used to compare the 12-month survival probabilities across ICI groups. The null hypothesis was that the survival probabilities were equal; Test type: Other; p = 0.289, Klein Method

7. Secondary Outcome: Local Control
Description: Local control was defined as the rate of any new, recurrent, or progressing tumor as defined by Response Assessment in Neuro-oncology (RANO) criteria within the planning target volume. This measure details the estimated 6-month survival and associated 95% confidence interval from the Kaplan Meier method. The time from treatment start to local failure was calculated. Patients who did not experience local failure were censored at the date last known alive or at the date of death if they expired.
Time Frame: 6 months
Population: Includes patients evaluable for 6-month outcomes.
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | Reduced Dose Stereotactic Radiosurgery With Immunotherapy
Number analyzed (Participants) | 12
survival probability | 1.00 [1.00 to 1.00]

8. Secondary Outcome: Local Control
Description: Local control was defined as the rate of any new, recurrent, or progressing tumor as defined by Response Assessment in Neuro-oncology (RANO) criteria within the planning target volume. This measure details the estimated 12-month survival and associated 95% confidence interval from the Kaplan Meier method. The time from treatment start to local failure was calculated. Patients who did not experience local failure were censored at the date last known alive or at the date of death if they expired.
Time Frame: 12 months
Population: Includes patients evaluable for 12-month outcomes.
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | Reduced Dose Stereotactic Radiosurgery With Immunotherapy
Number analyzed (Participants) | 12
survival probability | 0.913 [0.524 to 0.987]

9. Secondary Outcome: Local Control by SRS Group
Description: as for outcome 8
Time Frame: 12 months
Population: Includes patients who were evaluable for the 12-month outcomes.
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | Gamma Knife | Linear Accelerator
Number analyzed (Participants) | 8 | 4
survival probability | 1.00 [1.00 to 1.00] | 0.750 [0.128 to 0.961]
Statistical Analysis 1: Comparison: Gamma Knife vs Linear Accelerator; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.248, Klein Method

10. Secondary Outcome: Local Control by Brain Metastases Group
Description: as for outcome 8
Time Frame: 12 months
Population: Includes patients who were evaluable for the 12-month outcomes.
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | Melanoma Brain Metastases | Non-Melanoma Brain Metastases
Number analyzed (Participants) | 2 | 10
survival probability | 1.00 [1.00 to 1.00] | 0.900 [0.473 to 0.985]
Statistical Analysis 1: Comparison: Melanoma Brain Metastases vs Non-Melanoma Brain Metastases; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.292, Klein Method

11. Secondary Outcome: Local Control by Immune Checkpoint Inhibitor (ICI) Group
Description: as for outcome 8
Time Frame: 12 months
Population: Includes patients who were evaluable for the 12-month outcomes.
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | Single-Agent ICI | Multi-Agent ICI
Number analyzed (Participants) | 9 | 3
survival probability | 0.889 [0.433 to 0.984] | 1.00 [1.00 to 1.00]
Statistical Analysis 1: Comparison: Single-Agent ICI vs Multi-Agent ICI; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.289, Klein Method

12. Secondary Outcome: Radiographic Radiation Necrosis Rate
Description: Radiographic radiation necrosis was defined as brain imaging findings on magnetic resonance imaging (MRI), magnetic resonance (MR) perfusion, MR Spectroscopy, and/or positron emission tomography (PET) imaging consistent with radiation necrosis. This measure details the estimated 6-month survival and associated 95% confidence interval from the Kaplan Meier method. The time from treatment start to the presence of radiographic radiation necrosis was calculated. Patients who did not experience the outcome were censored at the date last known alive or at the date of death if they expired.
Time Frame: 6 months
Population: Includes the patients who were evaluable for the 6-month outcomes.
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | Reduced Dose Stereotactic Radiosurgery With Immunotherapy
Number analyzed (Participants) | 12
survival probability | 0.818 [0.447 to 0.951]

13. Secondary Outcome: Radiographic Radiation Necrosis Rate
Description: as for outcome 12
Time Frame: 12 months
Population: Includes the patients who were evaluable for the 12-month outcomes.
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | Reduced Dose Stereotactic Radiosurgery With Immunotherapy
Number analyzed (Participants) | 12
survival probability | 0.818 [0.447 to 0.951]

ADVERSE EVENTS:
Time Frame: Up to 28 Months
Description: Adverse events reported are those that are related to the SRS treatment and are as of February 2024. Patients are still on follow-up for the study and treatment-related adverse events can still occur. Patients were considered at risk for an adverse event if they started SRS treatment. For all-cause mortality and serious adverse events, treatment attribution was not considered.
Arm/Group | Reduced Dose Stereotactic Radiosurgery With Immunotherapy
All-Cause Mortality (participants affected / at risk) | 1/18
Serious Adverse Events (participants affected / at risk) | 1/18
Other Adverse Events (participants affected / at risk) | 7/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reduced Dose Stereotactic Radiosurgery With Immunotherapy (N=18)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Reduced Dose Stereotactic Radiosurgery With Immunotherapy (N=18)
Fatigue (General disorders) | 2
Headache (Nervous system disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-10): https://cdn.clinicaltrials.gov/large-docs/02/NCT04047602/Prot_SAP_000.pdf